CLINICAL TRIAL: NCT02684617
Title: Phase Ib Trial of Pembrolizumab (MK-3475) in Combination With Dinaciclib (MK-7965) in Subjects With Hematologic Malignancies (KEYNOTE-155).
Brief Title: Study of Pembrolizumab (MK-3475) in Combination With Dinaciclib (MK-7965) in Hematologic Malignancies (MK-3475-155/KEYNOTE-155)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-155; MK-3475-155 (Other: Merck Protocol Number); KEYNOTE-155 (Other: Merck)
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: rrCLL; rrMM; rrDLBCL
MeSH Terms: interventions — pembrolizumab; dinaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- rrCLL Cohort (Experimental): Participants with refractory chronic lymphocytic leukemia (rrCLL) received an infusion of pembrolizumab 200 mg followed by infusion of dinaciclib 7 mg/m^2 on Cycle 1 Day 1, and infusion of dinaciclib 10 mg/m^2 alone on Cycle 1 Day 8. Participants then received an infusion of pembrolizumab 200 mg followed by infusion of dinaciclib 14 mg/m^2 on Cycles 2-35 Day 1 and infusion of dinaciclib 14 mg/m^2 alone on Cycles 2-35 Day 8. Each cycle is 21 days.
  Interventions: Biological: pembrolizumab; Drug: dinaciclib
- rrMM Cohort (Experimental): Participants with relapsed or refractory multiple myeloma (rrMM) received an infusion of pembrolizumab 200 mg followed by infusion of dinaciclib 7 mg/m^2 on Cycle 1 Day 1, and infusion of dinaciclib 10 mg/m^2 alone on Cycle 1 Day 8. Participants then received an infusion of pembrolizumab 200 mg followed by infusion of dinaciclib 14 mg/m^2 on Cycles 2-35 Day 1 and infusion of dinaciclib 14 mg/m^2 alone on Cycles 2-35 Day 8. Each cycle is 21 days.
  Interventions: Biological: pembrolizumab; Drug: dinaciclib
- rrDLBCL Cohort (Experimental): Participants with relapsed or refractory diffuse large B-cell lymphoma (rrDLBCL) received an infusion of pembrolizumab 200 mg followed by infusion of dinaciclib 7 mg/m^2 on Cycle 1 Day 1, and infusion of dinaciclib 10 mg/m^2 alone on Cycle 1 Day 8. Participants then received an infusion of pembrolizumab 200 mg followed by infusion of dinaciclib 14 mg/m^2 on Cycles 2-35 Day 1 and infusion of dinaciclib 14 mg/m^2 alone on Cycles 2-35 Day 8. Each cycle is 21 days.
  Interventions: Biological: pembrolizumab; Drug: dinaciclib

INTERVENTIONS:
Biological: pembrolizumab — 200 mg administered as an intravenous (IV) infusion on Day 1 of infusion Cycles 1-35. Each cycle is 21 days.
  Other Names: MK-3475; SCH 9000475; KEYTRUDA®
Drug: dinaciclib — dinaciclib 7 mg/m^2 administered as an IV infusion on Day 1 of infusion Cycle 1, dinaciclib 10 mg/m^2 administered as an IV infusion on Day 8 of infusion Cycle 1, dinaciclib 14 mg/m^2 administered as an IV infusion on Days 1 and 8 of infusion Cycles 2-35. Each cycle is 21 days.
  Other Names: MK-7965

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pembrolizumab (MK-3475) used in combination with dinaciclib (MK-7965) in the treatment of relapsed or refractory chronic lymphocytic leukemia (rrCLL), multiple myeloma (rrMM), or diffuse large B-cell lymphoma (rrDLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Females must not be pregnant (negative urine or serum human chorionic gonadotropin test within 72 hours of study start)
* Female and male participants of reproductive potential must agree to use adequate contraception starting from the first dose of study medication, throughout the study period, and for up to 120 days after the last dose of study medication
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Cardiac function suitable for protocol-required hydration as determined by the investigator and/or cardiologist
* Must be able to provide biopsy specimens obtained ≤3 months for biomarker analysis. If bone marrow biopsy was performed 3 months before screening but subject had anti-cancer treatment after biopsy, the bone marrow biopsy and aspiration should be repeated

Relapsed or refractory chronic lymphocytic leukemia (rrCLL) participants:

* Must have a confirmed diagnosis of CLL defined by 2008 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
* Must have received one prior therapy for CLL
* Must meet one or more of the consensus criteria for initiating treatment

Relapsed or refractory multiple myelolma (rrMM) participants:

* Must have a confirmed diagnosis of active MM
* Must have undergone prior treatment with ≥2 treatment lines of anti-myeloma therapy and failed last line of treatment (disease progression ≤60 days of completion of last therapy)
* Must have failed prior anti-myeloma treatments that have included an immunomodulatory drug (IMiD) (pomalidomide, lenalidomide, or thalidomide) AND proteasome inhibitor (bortezomib, carfilzomib, or ixazomib) alone or in combination

Diffuse large B-cell lymphoma (rrDLBCL) participants:

* Must have a confirmed diagnosis of DLBCL and have progressed following ≥2 lines of previous therapy, after autologous stem cell transplant, or not a candidate for autologous stem cell transplant
* Must have measurable disease (≥1 lesion that is >15 mm in the longest diameter or by >10 mm in the short axis)

Exclusion Criteria:

* Has been treated with a cytochrome P450 3A4 (CYP3A4) strong inhibitor or inducer within 7 days of enrollment
* Has been treated with anti-cancer therapy or thoracic radiation therapy within 14 days
* Has known clinically active central nervous system (CNS) involvement
* Has a known history of immunosuppression or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days
* Has had prior anti-cancer monoclonal antibody within 4 weeks of Study Day 1 or who has not recovered from adverse events due to agents administered >4 weeks earlier
* Has undergone prior allogeneic hematopoetic stem cell transplantation within the last 5 years
* Has a known additional malignancy that is progressing or requires active treatment
* Has active autoimmune disease that has required systemic treatment in past 2 years
* Has an active infection requiring intravenous systemic therapy
* Has received prior therapy with an anti-programmed cell death-1 (PD-1), anti-programmed cell death ligand (PD-L) 1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) or chimeric antigen receptor (CAR)-T cell therapy or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has been previously treated with a cyclin-dependent kinase (CDK) inhibitor
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has a known history of or is positive for hepatitis B (hepatitis B surface antigen reactive) or hepatitis C (hepatitis C virus RNA [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has known current symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Relapsed or refractory chronic lymphocytic leukemia (rrCLL) participants:

* Has Richter's Transformation

Relapsed or refractory multiple myelolma (rrMM) participants:

* Participants with non-secretory or oligo-secretory myeloma, plasma cell leukemia or Waldenström's macroglobulinemia
* History of primary amyloidosis, hyperviscosity or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)

Diffuse large B-cell lymphoma (rrDLBCL) participants:

* Participants with primary mediastinal B-cell lymphoma (PMBCL)
* Has Richter's Transformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gregory GP, Kumar S, Wang D, Mahadevan D, Walker P, Wagner-Johnston N, Escobar C, Bannerji R, Bhutani D, Chang J, Hernandez-Ilizaliturri FJ, Klein A, Pagel JM, Rybka W, Yee AJ, Mohrbacher A, Huang M, Farooqui M, Marinello P, Quach H. Pembrolizumab plus dinaciclib in patients with hematologic malignancies: the phase 1b KEYNOTE-155 study. Blood Adv. 2022 Feb 22;6(4):1232-1242. doi: 10.1182/bloodadvances.2021005872. PMID 34972202
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The rrMM Cohort was closed to enrollment on 07-AUG-2017 due to lack of efficacy.
  The rrCLL Cohort was closed to enrollment on 30-APR-2019 due to lack of efficacy.
Period: Overall Study
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Started | 18 | 17 | 40
Treated | 17 | 17 | 38
Completed | 0 | 0 | 0
Not Completed | 18 | 17 | 40
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Death | 8 | 16 | 28
Not completed — Withdrawal by Subject | 2 | 0 | 4
Not completed — Screen Failure | 1 | 0 | 2
Not completed — Study Terminated by Sponsor | 6 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort | Total
Number analyzed (Participants) | 17 | 17 | 38 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (10.9) | 60.8 (9.5) | 64.1 (11.1) | 64.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 15 | 29
  Male | 14 | 6 | 23 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 4 | 5
  Not Hispanic or Latino | 17 | 16 | 34 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 16 | 14 | 32 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLTs consisted of the following if observed during treatment Cycles 1 or 2 and assessed by investigator to be possibly, probably, or definitely related to pembrolizumab or dinaciclib: grade 4 non-laboratory nonhematologic toxicity; grade 4 hematologic toxicity lasting >7 days (except thrombocytopenia); grade 4 thrombocytopenia of any duration; grade 3 thrombocytopenia if associated with bleeding; any grade 3 non-laboratory nonhematologic toxicity, except grade 3 nausea, vomiting, or diarrhea, which was not considered a DLT unless lasting more than 3 days despite optimal supportive care; Grade 3 or Grade 4 nonhematologic laboratory abnormality that required medical intervention, led to hospitalization, or persisted for >1 week; grade 3 or 4 febrile neutropenia; any drug-related AE that caused participant to discontinue treatment during Cycles 1 or 2; grade 5 toxicity; treatment-related toxicity that caused a >2-week delay in initiation of treatment Cycle 2 or 3. Each cycle was 21 days.
Time Frame: Up to 42 days
Population: The analysis population included all participants who received ≥1 dose of study medication, and who did not discontinue within the first two 21-day cycles of treatment or who experienced a DLT prior to completing the first two cycles of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 3 | 3 | 6
Participants | 1 | 1 | 1

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE was presented.
Time Frame: Up to approximately 582 days
Population: The analysis population included all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 17 | 17 | 38
Participants | 17 | 16 | 37

3. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study drug due to an adverse event is presented.
Time Frame: Up to 492 days
Population: The analysis population included all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 17 | 17 | 38
Participants | 4 | 2 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined in participants with CLL as the percentage of participants who have a confirmed Complete Response (CR) or Partial Response (PR) per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines (2008) as assessed by the investigator; in participants with DLBCL as the above definition but per the Revised Response Criteria for Malignant Lymphoma (2007) as assessed by the investigator; and in participants with MM as the percentage of participants who have a confirmed Stringent Complete Response (sCR), CR, PR, or Very Good Partial Remission (VGPR) per the International Uniform Response Criteria for Multiple Myeloma (2006) as assessed by the investigator.
Time Frame: Up to approximately 26 months
Population: The analysis population included all participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 17 | 17 | 38
Percentage of Participants | 29.4 [10.3 to 56.0] | 0.0 [0.0 to 19.5] | 21.1 [9.6 to 37.3]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the time from initial response to Progressive Disease (PD) or death, whichever occurred first. A response was: in participants with CLL, a confirmed Complete Response (CR) or Partial Response (PR) per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines (2008); in participants with DLBCL, as above but per the Revised Response Criteria for Malignant Lymphoma (2007); and in participants with MM, a confirmed Stringent Complete Response (sCR), CR, PR, or Very Good Partial Remission (VGPR) per the International Uniform Response Criteria for Multiple Myeloma (2006). The above guidelines also define PD by disease. Assessments were by investigator. Data were censored at last disease assessment documenting absence of PD for participants who: had no PD and were still on the trial; received antitumor treatment other than that of the trial; or were removed from trial prior to PD. DOR was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 26 months
Population: The analysis population included all participants who received ≥1 dose of study treatment and experienced a response to study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 5 | 0 | 8
Months | NA [NA to 11.1] — NA=Median DOR/DOR lower limit not reached |  | 4.9 [2.1 to NA] — NA=DOR upper limit not reached

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. PD evaluations were done based on the cancer-specific criteria of: the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines (2008) in participants with CLL; the Revised Response Criteria for Malignant Lymphoma (2007) in participants with DLBCL; and the International Uniform Response Criteria for Multiple Myeloma (2006) in participants with MM. Assessments were by investigator. PFS data were censored for participants with no PD or death at their last disease assessment, or at their last disease assessment prior to starting new anticancer treatment for those who did so. PFS was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 26 months
Population: The analysis population included all participants who received ≥1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 17 | 17 | 38
Months | 5.2 [1.4 to 12.4] | 1.6 [0.7 to 2.8] | 2.1 [1.8 to 2.6]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study treatment to death due to any cause. Data were censored at the date of a participant's last follow-up. OS was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who received ≥1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
Number analyzed (Participants) | 17 | 17 | 38
Months | 21.7 [9.5 to NA] — NA=OS upper limit not reached | 10.5 [2.6 to 13.5] | 7.9 [3.2 to 14.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 522 days for non-serious adverse events. Up to approximately 582 days for serious adverse events. Up to approximately 610 days for all-cause mortality.
Description: MedDRA preferred terms "neoplasm progression", "malignant neoplasm progression" and "disease progression" not related to the drug are excluded.
Arm/Group | rrCLL Cohort | rrMM Cohort | rrDLBCL Cohort
All-Cause Mortality (participants affected / at risk) | 9/17 | 16/17 | 32/38
Serious Adverse Events (participants affected / at risk) | 13/17 | 6/17 | 17/38
Other Adverse Events (participants affected / at risk) | 17/17 | 16/17 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rrCLL Cohort (N=17) | rrMM Cohort (N=17) | rrDLBCL Cohort (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (4) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rrCLL Cohort (N=17) | rrMM Cohort (N=17) | rrDLBCL Cohort (N=38)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 6 (6) | 6 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (13) | 2 (2) | 4 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (3) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 14 (19)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 10 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (10) | 4 (4) | 15 (18)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 4 (5)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 1 (2)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (3)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (12) | 6 (7) | 12 (15)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 8 (10)
Pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 7 (11)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (14)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (9) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Body height decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 2 (2) | 8 (11)
Lymphocyte count increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (7) | 0 (0) | 7 (9)
Platelet count decreased (Investigations) | 4 (4) | 4 (4) | 8 (8)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 6 (8)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 7 (8)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 6 (11)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 3 (3)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 5 (6)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 8 (8)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT02684617/Prot_SAP_000.pdf